CLINICAL TRIAL: NCT06725745
Title: Assessing Patient Centered Urological Care for Spina Bifida: a Collaboration Between the EAU-ESPU Pediatric Urology Guidelines Panel and the IFSBH.
Brief Title: A Collaboration Between the EAU-ESPU Pediatric Urology Guidelines and the IFSBH
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Lisette 't Hoen, Principal Investigator, Erasmus Medical Center
Other Study IDs: EMCSophia1
Record Dates: First submitted 2024-12-04; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Spina Bifida
Keywords: patient involvement; organization of care
MeSH Terms: conditions — Spinal Dysraphism; Patient Participation | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People with spina bifida: People with spina bifida are approached through representative organizations by email to complete a digital survey at 1 timepoint.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Survey containing a primary survey regarding basic demographic features, medical treatment and organization of care and two validated questionnaires.

SUMMARY:
Children with spina bifida require care from various medical and paramedical specialists throughout their life. The availability and organization of the care needed differs between the European countries. The EAU and IFSBH are both organizations with the aim to improve patient care and clinical outcomes for children with spina bifida.

The investigators have set up a collaboration to evaluate the differences in organization of care and clinical treatment received and how this affects outcomes with regard to quality of life and sexuality.

A digital survey has been constructed which will be distributed among children and adolescents with spina bifida and their caregivers. The IFSBH and national patient organizations will send out invitations to their members. Children and adolescents from 8 - 18 years of age with spina bifida are eligible for inclusion.

The survey includes a primary survey developed in collaboration between panel members of the EAU pediatric urology guidelines and patient representatives. The second part includes validated questionnaires to evaluate Quality of life with the QUALAS and sexual function with the IIEF-5/FSFI-6 for boys/girls respectively.

Primary outcome will be the quality of life in children and adolescents with spina bifida. The team will evaluate if their demographic differences influence the quality of life and if differences are seen between the different European countries. Secondary outcomes include differences in sexual function, organization of care, treatment received, treatment options available, with also a focus on differences between the different European countries.

The results of this survey will be evaluated and interpreted within a sounding board group consisting of children/adolescents/adults with spina bifida, patient representatives from IFSBH and panel members of the EAU Pediatric Urology guidelines panel. Finally, the interpreted results will be used to update the EAU Pediatric Urology guidelines to make these more patient centered.

There are no known risks of participating in the study given the fact that participation includes only completion of questionnaires and data about standard of care. Furthermore, the study is completely voluntary and the results will be completely anonymous.

DETAILED DESCRIPTION:
Introduction and rationale Children with spina bifida require care from various medical and paramedical specialists throughout their life. The availability and organization of the care needed differs between the European countries. It can be expected that this variety results in differences in outcome of care.

Children with spina bifida have stated that for future research they feel it is important that quality of life and sexuality are investigated.

The EAU Pediatric Urology guidelines panel wants to ensure that patients with spina bifida receive the best possible care based on the best available clinical evidence. Additionally, this team wants to improve the clinical guidelines by including patients perspectives. The IFSBH represents patients with spina bifida and values the promotion and protection of the human rights of patients with spina bifida thereby improving quality of life.

Together with the IFSBH the investigators have set up a collaboration to investigate how the team can make the guidelines more patient centered and thereby improve quality of care and quality of life.

For this aim the investigators have developed a survey to evaluate the current organization of care, demographic features and received treatment. The outcome of this survey will show the exact differences in care between European countries. The investigators have included two validated questionnaires to measure the effect this has on quality of life and sexuality. The information gathered will be used to adapt the clinical EAU Pediatric Urology guidelines.

Objective(s) The main objective is to improve the quality of life of patients with spina bifida by updating the guidelines according to the differences found in care and how this impacts patients outcomes.

The team will evaluate the difference in organization of care between different European countries based on the outcomes of the primary survey. The baseline quality of life and sexuality reported will be evaluated with the QUALAS and the IIEF-5/FSFI-6 questionnaires. The investigators will then explore the relationship between how care is organized and how this affects quality of life and sexuality. The results of this study will be used to update the EAU Pediatric Urology clinical guidelines. Also, it will highlight the direction for future research to improve patients care and thereby quality of life and/or sexuality, which patients with spina bifida have stated they themselves find important.

Methods This digital survey includes a primary survey regarding basic demographic features, medical treatment and organization of care. This survey was constructed by the EAU guidelines panel and the IFSBH patient representatives. The second part of the digital survey includes two validated questionnaires. The QUALAS is a validated questionnaire regarding quality of life in patients with spina bifida. There are two different versions for the ages 8-12 and 13-18 years. To evaluate sexuality the IIEF-5 (for boys) and the FSFI-6 (for girls) are used. These questionnaires are validated and are used in patients with spina bifida to evaluate sexual function as standard of care. Only children aged 13 years or older will be asked if they want to answer questions about sexuality and if they answer yes they will be asked for which gender they want to answer questions about their sexuality. After this they'll get the IIEF-5 or FSFI-6 questionnaire.

This digital survey is available in nine languages: English, Spanish, German, Italian, French, Danish, Greek, Turkish and Dutch.

The link to surveymonkey will be distributed by the IFSBH and local patient organizations among their members.

After the data have been collected, the general results of the survey will be evaluated and interpreted with a sounding board group. When patients participate with the digital survey they will not be involved in the sounding group. This sounding board group will consist of children/adolescents/adults with spina bifida who are representatives from the patient organization IFSBH and panel members of the EAU. This sounding board group will meet for a day. Finally, the results will be used to update the EAU Pediatric Urology guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Must have spina bifida
* Must be able to complete the digital survey, with help of caregivers allowed.
* Speak one of the nine available languages:

  * English,
  * Spanish,
  * German,
  * Italian,
  * French,
  * Danish,
  * Greek,
  * Turkish,
  * Dutch

Exclusion Criteria:

* Does not have spina bifida

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with spina bifida who are approached by their representative organizations
Sampling Method: Probability Sample
Enrollment: 281 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
QUALAS score | 6 months
  Score derived from the Quality of Life Assessment in Spina Bifida (QUALAS) survey Scores range from 0-100 with higher scores indicating better quality of life

SECONDARY OUTCOMES:
Demographic parameters | 6 months
  Gender, age, medication use, catheter use, organization of care
IIEF score | 6 months
  Score derived from the International Index of Erectile Function (IIEF) survey Scores range from 1-25 with higher scores indicating better erectile function
FSFI score | 6 months
  Score derived from the Female Sexual Function Index (FSFI) survey. Scores range from 2-30 with higher scores indicating better sexual function

CONTACTS AND LOCATIONS:
Overall Officials: Lisette 't Hoen, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-15): https://cdn.clinicaltrials.gov/large-docs/45/NCT06725745/Prot_SAP_000.pdf